CLINICAL TRIAL: NCT00620984
Title: Staphylococcus Aureus Carrier Status in Breastfeeding Mothers and Infants and the Risk of Lactation Mastitis: A Large Prospective Study
Brief Title: Staphylococcus Aureus Carrier Status in Breastfeeding Mothers and Infants and the Risk of Lactation Mastitis
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Jayne Charlamb, MD, Assistant Professor of Obstetrics and Gynecology, State University of New York - Upstate Medical University
Other Study IDs: 5395
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Mastitis; Staphylococcus Aureus; Staphylococcal Infections
Keywords: Staphylococcus aureus; Breastfeeding; Lactational Mastitis; Polymerase Chain Reaction (PCR) amplification analysis; staphylococcal infections; staphylococcal Carrier State
MeSH Terms: conditions — Mastitis; Staphylococcal Infections; Breast Feeding; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Lactation (breastfeeding) mastitis is an acute infection of the milk ducts of the breastfeeding woman. Staphylococcus aureus (S. aureus) is the infectious germ most commonly associated with lactation mastitis. Twenty percent of the general population are carriers of Staphylococcus aureus, which means that they carry the infectious germ but do not become ill from it. It has been suggested that mothers who are carriers of S. aureus in their nostril may be at an increased risk of developing lactational mastitis, however; this has not been clinical proven.

We are studying the relationship between S. aureus carrier status of breastfeeding mothers and infants and the risk of developing lactational mastitis. Additionally, we are collecting questionnaire data in an attempt to better define factors predisposing women to lactation mastitis.

DETAILED DESCRIPTION:
Lactation mastitis is an acute inflammation of the interlobular connective tissue within the mammary gland of a breastfeeding woman. It is a relatively common condition that causes pain and worry, and can lead to restriction in activity and increased risk of early weaning from breastfeeding. Staphylococcus aureus is the infectious agent most commonly implicated in lactation mastitis.

It is well established that the anterior nares are the primary reservoir of S. aureus in humans and that approximately 20% of healthy individuals are "persistent carriers" of the organism. Carriage of Staphylococcus aureus has been identified as a significant risk factor for the development of infection including surgical wound infections. It has been suggested that maternal and infant nasal carriage of S. aureus may be associated with an increased risk of breast infection during lactation.

We propose to prospectively study the relationship between the S. aureus carrier status of 500 healthy breastfeeding dyads and the rate of the subsequent development of lactational mastitis. Carrier status of mothers and infants will be determined through two nasal swabbings performed in the early post-partum period. The swabs will be analyzed with both traditional culture and through Polymerase chain reaction (PCR) amplification analysis. Mastitis rate will be determined via serial follow-up telephone interviews during the first two months post-partum.

ELIGIBILITY:
Inclusion Criteria:

* Mother must plan to breastfeed exclusively for at least two months
* Mother must be 18 years or older.
* Mother must speak English and capable of giving informed consent
* Must be the delivery of a term (37 weeks or more), singleton live infant.
* Mother must be within post-partum day zero to three-status post delivery
* Both mother and infant generally healthy without disease known to cause significant immune dysfunction or known to be associated with abnormally high carriage rates of S. aureus such as HIV-positive status or AIDS, Type I Diabetes Mellitus, ongoing need for hemodialysis or chronic steroid use, or receiving either chemotherapy/radiation treatment for malignancy?
* Must have the ability to communicate via phone for follow up assessments.

Exclusion Criteria:

* Does not have the ability to drop off the second set of cultures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will be enrolling 500 dyads (mother and newborn infant pairs) into the study over approximately a three year period. Mothers will be age 18 years or older.
Sampling Method: Probability Sample
Enrollment: 557 (Actual)
Dates: Start 2006-08; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Our primary objective is to determine the association of nasal carriage of S. aureus in breastfeeding mothers and infants with the rate development of mastitis in the mothers. | Culture results will be unblinded at the end of the study.

SECONDARY OUTCOMES:
Secondary objective will be to document the S. aureus carriage rate, including methicillin-resistant Staphylococcus aureus (MRSA), in early post-partum period and to assess the relationship between S. aureus carrier status of the mother and the infant. | Culture results will be unblinded at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jayne R Charlamb, MD, IBCLC, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States